CLINICAL TRIAL: NCT02741934
Title: Cognitive and Behavioral Outcomes of School-aged Children Who Were Born Preterm
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: KangWon National University Hospital (Other)
Responsible Party: Principal Investigator, Ee-Kyung Kim, Clinical associate professor, Seoul National University Hospital
Other Study IDs: 2015-1927
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Very Low Birth Weight Infants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Preterm cohort: Among the infants who were born and admitted to Seoul National University Hospital from 2008 to 2009, the birth weight of the infants less than 1,500g or gestational age less than 32 weeks patients were enrolled.
- Term control cohort: The infants who were born from 2008 to 2009 with term gestational age will be enrolled.

SUMMARY:
This study evaluates the cognitive and behavioral outcomes including image findings of school-aged children who were born preterm compared with who were born term gestational age.

DETAILED DESCRIPTION:
There are lots of studies published that school-aged children who were born preterm has some behavioral problems in school and they also have poor academical achievement.

ELIGIBILITY:
Inclusion Criteria:

* children former preterm infants < 32 weeks of gestation or 1,500gm of birth weight
* children former normal term infants

Exclusion Criteria:

* major congenital anomaly
* neuromuscular disease
* chromosomal anomaly

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Among the infants who were born and admitted to Seoul National University Hospital from 2008 to 2009, the birth weight of the infants less than 1,500g or gestational age less than 32 weeks patients were enrolled.
  The infants who were born from 2008 to 2009 with term gestational age will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cognitive function test | 8 Years old

SECONDARY OUTCOMES:
Brain MRI | 8 Years old
Korean Child Behavior Checklist | 8 Years old
Korean ADHD Rating Scale-IV | 8 Years old
Wechsler Scale of Intelligence-IV | 8 Years old
Advanced Test of Attention | 8 Years old
Children's color trails test | 8 Years old
STROOP | 8 Years old
Wisconsin Card Sorting Test | 8 Years old

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No